CLINICAL TRIAL: NCT01163474
Title: Telemedicine in Cardiac Surgery: A Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PPO 10-060
Record Dates: First submitted 2010-07-14; First posted 2010-07-15 (Estimated); Results first posted 2015-01-05 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Coronary Artery Disease
Keywords: Telemedicine; Surgery, Cardiac
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 - All study participants (Experimental): Evaluate video clinic visit prior to Face-to-Face usual care visit
  Interventions: Other: Evaluate video clinic visit prior to Face-to-Face usual care visit

INTERVENTIONS:
Other: Evaluate video clinic visit prior to Face-to-Face usual care visit — Evaluate video clinic visit prior to Face-to-Face usual care visit
  Other Names: video teleconference visit

SUMMARY:
Telemedicine has been widely used in managing patients with neurologic disorders or mental illness. Telemedicine is defined as the use of medical information exchanged from one site to another via electronic communications for the health and education of the patient or healthcare provider and for the purpose of improving patient care. According to our knowledge, it has not been used to manage cardiac patients who need postoperative care after discharge from hospitals.

The use of telemedicine has the potential to reduce the cost of unnecessary travel by assessing the patient's postoperative status prior to making decisions as to whether or not a face-to-face consultation is necessary.

In this pilot study we will compare the accuracy of surgeons' decisions during follow-up visits via video-teleconference (V-Visit) to surgeons' decisions during traditional face-to-face follow-up visits (FTF-Visits). Both the V-Visit and the FTF-Visit will take place at the Houston Michael E DeBakey VA Medical Center on the same day. We will also ask both patients and providers to complete short questionnaires after each V-Visit regarding their acceptability of using telemedicine for these post-operative follow-up visits.

Information collected as part of this pilot study will be used to design a future full randomized controlled trial (RCT) on the use of telemedicine in evaluating post-operative cardiac surgical patients.

DETAILED DESCRIPTION:
The specific aims are:

1. To compare surgeons' decisions on patient disposition between V-visits and FTF-visits (gold standard).
2. To assess the acceptability to patients and surgeons of using V-visits in the postoperative care of cardiac surgical patients;
3. To assess the technical feasibility of using community-based outpatient clinics (CBOCs) for delivery of postoperative cardiac surgical care;
4. To determine the recruitment rate for eligible subjects.

We plan to conduct this pilot study at the Michael E. DeBakey Veterans Affairs Medical Center (MEDVAMC) in Houston, Texas, along with satellite CBOC facilities in Lufkin and Conroe. Once the accuracy, acceptability, and feasibility of the use of video conferencing (VC) in the postoperative care for cardiac surgical patients are established, we will submit a full proposal to conduct a two-arm RCT in future.

ELIGIBILITY:
Inclusion Criteria:

1. Patients older than 18 years of age
2. Patients who have undergone one of the following cardiac surgical procedures:

Coronary artery bypass grafting (CABG) and/or Cardiac valvular operations

Exclusion Criteria:

1. Patients who have undergone aortic dissection/aneurysm operations
2. Patients who have been diagnosed with atrial fibrillation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Danny Chu, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, TX, Houston, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited after coronary artery bypass or cardiac valvular surgery.
Pre-assignment Details: All participants were assigned to both the intervention (post-surgical evaluation by video-teleconference) and control (face-to-face visit) groups.
Groups:
- Arm 1 - Evaluate Video Clinic Visit Prior to Face-to-Face Usua: Evaluate video clinic visit prior to Face-to-Face usual care visit
Period: Overall Study
Arm/Group | Arm 1 - Evaluate Video Clinic Visit Prior to Face-to-Face Usua
Started | 40
Completed | 24
Not Completed | 16
Not completed — Withdrawal by Subject | 1
Not completed — Tech barriers to videoteleconference vis | 12
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 - Evaluate Video Clinic Visit: Evaluate video clinic visit prior to Face-to-Face usual care visit
Arm/Group | Arm 1 - Evaluate Video Clinic Visit
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 64 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24
Race/Ethnicity, Customized [Number; unit: participants]
  White | 16
  African American | 4
  Hispanic | 4
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Accuracy (FTF Decision on Patient Disposition vs. V-visit Decision on Patient Disposition)
Description: Using CVT software and desktop webcams on the VA private network, "Virtual" CVT visits were conducted immediately prior to usual care of Face-to-Face (FTF) postoperative visits. Two independent surgeons reviewed the CVT recordings and made recommendations on patient dispositions. Accuracy was assessed by comparing the 2 reviewers' CVT decisions to the FTF decision.
Time Frame: 1 month
Measure: Number; unit: percentage of agreement
Groups:
- Arm 1 - Evaluate Video Conferencing: Evaluate virtual video conference follow-up clinic visit
  Evaluative process: Evaluative process using video conferencing
Arm/Group | Arm 1 - Evaluate Video Conferencing
Number analyzed (Participants) | 24
percentage of agreement | 89

2. Secondary Outcome: Acceptability
Description: Acceptability was assessed using a the Demeris 17-item Likert-scale questionnaire. Scale from 1 to 5 (1 = strongly disagree; 5 = strongly agree).
Time Frame: 1 month
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm 1 - Provider Evaluate Video Conferencing: Evaluate virtual video conference follow-up clinic visit
  Evaluative process: Evaluative process using video conferencing
Arm/Group | Arm 1 - Provider Evaluate Video Conferencing
Number analyzed (Participants) | 23
units on a scale | 68 (6.7)

3. Secondary Outcome: Feasibility
Time Frame: 1 month
Population: Data for this outcome are no longer available.
Arm/Group | Arm 1 - Evaluate Video Clinic Visit Prior to Face-to-Face Usua
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Arm 2: Face-to-face follow up for subjects (control)
Arm/Group | Arm 1 - Evaluate Video Conferencing | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 0/24 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes